CLINICAL TRIAL: NCT07194096
Title: Preoperative Stress Hyperglycemia Ratio and Postoperative Delirium
Brief Title: Stress Hyperglycemia Ratio and Postoperative Delirium
Status: Not yet recruiting | Type: Observational
Sponsor: Rao Sun (Other)
Responsible Party: Sponsor-Investigator, Rao Sun, Associate chief physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202509010A
Record Dates: First submitted 2025-09-05; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Postoperative delirium is a common and serious complication associated with prolonged hospitalization, increased morbidity and mortality, and elevated healthcare costs. Identifying reliable predictive biomarkers for early risk stratification is crucial for implementing preventive strategies and improving patient outcomes.

The stress hyperglycemia ratio (SHR) is an emerging biomarker that quantifies stress-induced hyperglycemia relative to baseline glycemic status, providing an assessment of physiological stress. This metric has been associated with various adverse outcomes. Given that surgical stress triggers neuroendocrine and inflammatory responses potentially contributing to delirium pathogenesis, SHR may indicate vulnerability to postoperative cognitive dysfunction.

The primary objective of this retrospective study is to investigate the association between preoperative stress hyperglycemia ratio and postoperative delirium development. Additionally, we aim to evaluate the predictive value of preoperative SHR for postoperative delirium risk stratification. This investigation may provide insights into metabolic stress-related mechanisms underlying postoperative cognitive outcomes and identify a clinically applicable biomarker for delirium risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Underwent non-neurosurgical and non-cardiac surgical procedures
* For patients with multiple qualifying surgical procedures during the study period, only data from the first eligible surgery were analyzed

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status V
* Procedural sedation or anesthesia performed outside the operating room, or total anesthesia duration ≤60 minutes
* Preoperative delirium or dementia
* Insufficient laboratory data for calculating the stress hyperglycemia ratio (SHR)
* Missing values for essential confounding variables required for multivariable analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years or older who underwent non-neurosurgical and non-cardiac surgical procedures at Tongji Hospital between 2014 and 2024 were included.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative delirium | Perioperative/Periprocedural

CONTACTS AND LOCATIONS:
Overall Officials: Rao Sun, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No